CLINICAL TRIAL: NCT06958731
Title: Out-of-plane Versus Real-time Bi-plane Single-operator Laser-assisted With a Innovative T-shaped Probe for Ultrasound-guided Internal Jugular Vein Catheterization: A Randomized Clinical Trial
Brief Title: To Compare the Success Rate of Internal Jugular Vein Catheterization at the First-attempt Between Single-operator Laser-assisted T-shaped Probe and Traditional Ultrasound-guided Out-of-plane Technique in Adults (≥ 18 Years of Age).
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25K114-001
Record Dates: First submitted 2025-04-20; First posted 2025-05-06 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2024-12

CONDITIONS: Patients Were Over 18 Years and Older Who Required IJVC

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the single-operator Laser-assisted T-shaped probe ultrasound-guidance group (Experimental)
  Interventions: Device: TuoRen Ultrasonic System
- traditional ultrasound-guided out-of-plane group (Experimental)
  Interventions: Device: Huasheng Color Ultrasonic Diagnostic System

INTERVENTIONS:
Device: TuoRen Ultrasonic System — The Single-operator Laser-assisted T-shaped probe consisted of TuoRen Ultrasonic System (TUR200, Shenzhen Tuoren Bio-Medical Electronics Co., LTD) with a T-shaped probe (L38T7C), a 3D-printed probe-carrying enclosure with a linear laser transmitter ( ZLM120AL650-22130BXS, Shenzhen Zhonglai Technology Co., Ltd.) and ultrasonic probe manipulator.
  Arms: the single-operator Laser-assisted T-shaped probe ultrasound-guidance group
Device: Huasheng Color Ultrasonic Diagnostic System — Ultrasonic (Huasheng Color Ultrasonic Diagnostic System, Navi s, Shenzhen Huasheng Medical Technology Co., LTD.) and a 4.0MHz phased probe were used for the short-axis out-of-plane internal jugular vein catheterization
  Arms: traditional ultrasound-guided out-of-plane group

SUMMARY:
Background: Ultrasound guidance is an important technique to improve the success rate of internal jugular vein catheterization (IJVC) at the first-attempt, however, both long-axis in-plane and short-axis out-of-plane techniques have their own disadvantages. The T-shaped ultrasonic probe invented by us combined with the help of laser positioning and 3D printing manipulator could realize real-time bi-plane guidance of the needle short-axis out-of -plane and long-axis in-plane. With the help of the Single-operator Laser-assisted T-shaped probe, the whole process of needle insertion, guide wire placement and catheter placement can be visualized, which is expected to improve the success rate on the first-attempt.

Objective: The primary outcome was the first-attempt success rate of RIJV catheterization. The completion of the catheterization was defined as the presentation of the CVP waveform on the monitor. The secondary outcomes included the first-attempt success rate of guidewire placement, the procedure time to success within the first-attempt, procedure time to success within the second attempt, overall procedure time, overall success rate, equipment preparation time, location time, number of unintentional penetration events of the posterior wall, average number of adjustments.

Design, Setting, and Participants: This single-center, prospective, parallel-group, randomized controlled study enrolled surgical patients over 18 years and older (ASA grade Ⅰ-Ⅲ) who required IJVC in the First Hospital of Jilin University. The exclusion criteria were prior puncture at the same site in the previous month; puncture site injury, infection, or hematoma; peripheral vascular disease; congenital heart disease, hypovolemia or cardiogenic shock, and severe arrhythmia. The participants were randomized into the traditional ultrasound-guidance group or the single-operator Laser-assisted T-shaped probe ultrasound-guidance group. After inducing general anesthesia, ultrasound-guided internal jugular vein catheterization was performed by two experienced operators.

Interventions: Patients were randomly assigned to undergo the Single-operator Laser-assisted T-shaped probe group (n = 54) or traditional ultrasound-guided group (n = 54).

Randomization and Trial Procedures: The randomization website (https://www.randomizer.org) was used by the research statistician to generate random unique numbers from 1 to 108, which were then sealed into opaque numbered envelopes with grouping information. The subjects were randomly assigned (1:1) to Single-operator Laser-assisted T-shaped probe group or traditional ultrasound-guided group. The operator team that was not involved in any other part of the study, consisted of doctor A and doctor B. These two residents should had participated in clinical work for more than five years and were proficient in the two ultrasound-assisted methods and successfully completed more than 50 cases of alone. In view of the notably different settings of the two techniques, the allocation was not blinded to the operators, equipment assistant, and research assistant. Conversely, the relatives of the subjects were blinded to the group assignment and free to withdraw from the trial at any time. All data were collected and analyzed by the same research assistant.

Statistical Analysis: The sample size required for this study was calculated using PASS 21.0 (NCSS, USA). According to a pilot study in our department, the success rate of the first attempt was 98% in the the T-shaped probe combined with laser group, and according to the relevant literature, the success rate of first-attempt in traditional ultrasound-guided group was 77%. Considering a dropout rate of 10%, the required sample size in the present study was 108 patients per group (two sided α = 0.05; power = 0.90).

Shapiro-wilk test was used to test the normality of measurement data. The measurement data with normal distribution were described by mean ± standard deviation, and the measurement data with non-normal distribution were described by median (lower quartile, upper quartile). Count data were described by frequency (percentage). Independent t-test, χ2 test were used to assess the baseline characteristics of the study population, and GLM analysis was used to adjust the effect of covariates; The main outcome measures were analyzed using the χ2 test. Secondary outcomes were analyzed using the chi-square test, Fisher's exact test and Mann-Whitney U test. All statistical analyses were performed using IBM SPSS Statistics 24 (SPSS Corporation, IBM Corporation, USA). Statistical significance was defined as a two-sided P-value of less than 0.05.

DETAILED DESCRIPTION:
The vital signs of the patients were monitored when entering the operating room. After the establishment of peripheral venous access, the patients received rapid induction of general anesthesia and tracheal intubation. Without special circumstances, the right internal jugular vein was selected by the operator after randomization. The probe frequency of 13 MHz and a depth of 4.0 cm were set for optimal image quality in both groups. The patient was placed in a supine position with the head 15 degrees lower and the head turned to the left to fully expose the right side of the neck, and a thin pillow was placed under the right shoulder if necessary. After hand sterilization, the operator disinfected the puncture site and the surrounding skin with iodophor. An aseptic surgical drape was laid subsequently. With the help of the equipment assistant applying the coupling agent on the surface of the ultrasound probe, the operator with sterile gloves tightly wrapped the device composed of the probe, the enclosure and manipulator with the sterile sheath. Sterile coupling agent was again applied outside of the sterile sheath after scattered air bubbles were completely extruded.

In the Single-operator Laser-assisted T-shaped probe group, before the patient entered the operation room, the assistant prepared the equipment with the laser emitter was fixed to the T-shaped probe. And the adjustable belt was fastened to ensure that the probe was more closely combined with the enclosure and the manipulator. Procedure for RIJV localization with T-shaped probe: Step 1: the T-shaped probe was placed at the level of the patient's thyroid cartilage, and the ultrasound midline of short axis passed through the middle of the RIJV's cross-section; the probe was fixed in this position by the manipulator to make the image clear, which improved the shortcomings of hand-held probe which caused venous deformation due to too large force or image loss due to too small force. Step 2: the long axis of the ultrasound probe was fan-shaped to swing from side to side with the midline of the short axis of the T-shaped probe as the circle center until the long axis image of the RIJV was clearly displayed (see red rectangle on sonogram at upper left, and the red dashed line indicates at the same depth) at the corresponding depth with the RIJV on the short axis. Side view of schematic diagram of RIJV location: the vessel covered below the T-shaped probe is the puncture target vessel, while the laser can be considered as the surface navigation in the direction of the target vessel. After the assistant helped turn on the laser source, the operator held the needle in his right hand and allowed the laser beam to completely cover the needle so that the needle direction is right perpendicular to the short axis of target RIJV. Eventually, the height of the ultrasonic screen was lowered to the operator's eye level to reduce head-neck movements in favor of guiding convenience. For the traditional ultrasound-guided short-axis out-of-plane group, all preparation procedures were repeated as described in the ultrasound-guided short-axis out-of-plane technique.

ELIGIBILITY:
Inclusion Criteria:

* Undergo elective surgery
* Require internal jugular vein catheterization
* ASA grade I~Ⅲ
* Over 18 years and older

Exclusion Criteria:

* Prior puncture at the same site in the previous month
* Puncture site injury, infection, or hematoma
* Peripheral vascular disease
* Congenital heart disease, hypovolemia or cardiogenic shock, and severe arrhythmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
the first-attempt success rate | perioperative/periprocedural

SECONDARY OUTCOMES:
the first-attempt success rate of guidewire placement | perioperative/periprocedural
the procedure time to success within the first-attempt | perioperative/periprocedural
the procedure time to success within the second attempt | perioperative/periprocedural
the overall procedure time | perioperative/periprocedural
the overall success rate | perioperative/periprocedural
the equipment preparation time | perioperative/periprocedural
location time | perioperative/periprocedural
average number of adjustments | perioperative/periprocedural
complications | perioperative/periprocedural

CONTACTS AND LOCATIONS:
Locations (1):
- the first hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No